CLINICAL TRIAL: NCT02980341
Title: Phase 1/2, Multicenter, Open-label, Multiple-Dose First-in-human Study of U3-1402, in Subjects With HER3 Positive Metastatic Breast Cancer
Brief Title: Phase I/II Study of U3-1402 in Subjects With Human Epidermal Growth Factor Receptor 3 (HER3) Positive Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo Co., Ltd. (Industry)
Collaborators: Daiichi Sankyo (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: U31402-A-J101; JapicCTI-163401 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2016-11-28; First posted 2016-12-02 (Estimated); Results first posted 2024-08-13 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Oncology; HER3; Antibody drug conjugate; Developmental Phase I/II
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — patritumab deruxtecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Escalation Part (Experimental): Participants receive U3-1402 from 1.6 mg/kg to 8.0 mg/kg, administered via intravenous (IV) solution at 3-week intervals.
  Interventions: Drug: Patritumab Deruxtecan
- Dose Finding Part (Experimental): Participants receive 1 of 5 different U3-1402 dosing regimens, administered via IV solution at 2 or 3-week intervals at doses at or lower than those studied in the Dose Escalation Part.
  Interventions: Drug: Patritumab Deruxtecan
- Dose Expansion Part (Experimental): Participants with HER3 high, HER2 negative, HR positive status receive 4.8 mg/kg or 6.4 mg/kg of U3-1402 administered via intravenous (IV) solution at 3-week intervals. Participants with HER3 low, HER2 negative, HR positive status receive 6.4 mg/kg of U3-1402 administered via intravenous (IV) solution at 3-week intervals. Participants with HER3 high, HER2 negative, HR negative status receive 6.4 mg/kg of U3-1402 administration via intravenous (IV) solution at 3-week intervals.
  Interventions: Drug: Patritumab Deruxtecan

INTERVENTIONS:
Drug: Patritumab Deruxtecan — U3-1402 consists of an antibody component (patritumab, U3-1287) covalently conjugated to a drug-linker (MAAA-1162a) containing a drug component (MAAA-1181a)
  Other Names: U3-1402

SUMMARY:
This is an open-label, three-part, multiple-dose study to evaluate safety, tolerability, and efficacy of U3-1402 in patients with HER3-positive metastatic breast cancer. HER3 is a unique member of the human epidermal growth factor receptor, which defines a certain type of cancer.

The number of patients and treatment cycles are not fixed in this study. Subjects who continue to derive clinical benefit from the study treatment in the absence of withdrawal of consent, progressive disease (PD), unacceptable toxicity, or death may continue the study treatment until the end of the trial.

ELIGIBILITY:
Key Inclusion Criteria:

1. Is 18 Years and older in the United States or 20 Years and older in Japan
2. Has a pathologically documented advanced/unresectable or metastatic breast cancer
3. Documented HER3-positive disease measured by immunohistochemistry (IHC)
4. Has disease that is refractory to or intolerable with standard treatment, or for which standard treatment no longer is available
5. Has an Eastern Cooperative Oncology Group Performance Status 0-1
6. Has Left Ventricular Ejection Fraction ≥ 50%
7. Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

   Additional Inclusion Criteria for Dose Finding Part and Dose Expansion Part:
8. Has received 2-6 prior chemotherapy regimens for breast cancer, at least 2 of which were administered for treatment of advanced/unresectable or metastatic disease. At least 1 prior chemotherapeutic regimen must have included a taxane, administered in the neoadjuvant, adjuvant, or advanced setting. (With exception of Dose Expansion Part TNBC cohort. See additional inclusion criteria for Dose Expansion Part TNBC cohort.)

   Additional Inclusion Criteria for Dose Expansion Part Only:
9. Is able to submit a fresh tumor biopsy sample prior to starting study treatment if not already submitted for HER3 expression
10. Has documented hormone (estrogen and/or progesterone) receptor (HR)-positive and HER2 negative expression according to American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines. (With exception of Dose Expansion Part TNBC cohort. See additional inclusion criteria for Dose Expansion Part TNBC cohort.)

    Additional Inclusion Criteria for Dose Expansion Part TNBC cohort Only:
11. Has documented hormone (estrogen and progesterone) receptor (HR)-negative and HER2 negative expression according to American Society of Clinical Oncology - College of American Pathologists (ASCO-CAP) guidelines
12. Has progressed after receiving 1 to 2 prior chemotherapy regimens for advanced/unresectable or metastatic breast cancer.

Key Exclusion Criteria:

1. Prior treatment with a HER3 antibody
2. Prior treatment with an antibody-drug conjugate (ADC) which consists of an exatecan derivative that is a topoisomerase I inhibitor (eg, DS-8201)
3. Has a medical history of symptomatic congestive heart failure (New York Heart Association classes II-IV) or serious cardiac arrhythmia requiring treatment
4. Has a medical history of myocardial infarction or unstable angina
5. Has a corrected QT prolongation to > 450 millisecond (ms) in males and > 470 ms in females
6. Has a medical history of clinically significant lung diseases (eg, interstitial pneumonia, pneumonitis, pulmonary fibrosis, and radiation pneumonitis) or who are suspected to have these diseases by imaging at screening period
7. Has clinically significant corneal disease

   Additional Exclusion Criteria for Dose Expansion Part:
8. Prior treatment with an govitecan derivative (eg, IMMU-132).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (26):
- United States (10):
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Texas Oncology, P.A., Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Mays Cancer Center, San Antonio, Texas
- Japan (16):
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - National Cancer Center Hospital East, Chiba
  - Fukushima Medical University Hospital, Fukushima
  - Local Independent Administrative Corporation Hiroshima City Hospital Organization Hiroshima City Hiroshima Citizens Hospital, Hiroshima
  - Hakuaikai Social Medical Corporation Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Aichi Cancer Center Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osaka
  - Saitama Medical University International Medical Center, Saitama
  - Saitama Cancer Center, Saitama
  - National Cancer Center Hospital, Tokyo
  - The Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/ .
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Krop IE, Masuda N, Mukohara T, Takahashi S, Nakayama T, Inoue K, Iwata H, Yamamoto Y, Alvarez RH, Toyama T, Takahashi M, Osaki A, Saji S, Sagara Y, O'Shaughnessy J, Ohwada S, Koyama K, Inoue T, Li L, Patel P, Mostillo J, Tanaka Y, Sternberg DW, Sellami D, Yonemori K. Patritumab Deruxtecan (HER3-DXd), a Human Epidermal Growth Factor Receptor 3-Directed Antibody-Drug Conjugate, in Patients With Previously Treated Human Epidermal Growth Factor Receptor 3-Expressing Metastatic Breast Cancer: A Multicenter, Phase I/II Trial. J Clin Oncol. 2023 Dec 20;41(36):5550-5560. doi: 10.1200/JCO.23.00882. Epub 2023 Oct 6. PMID 37801674

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 182 participants who met all inclusion criteria and no exclusion criteria received at least 1 dose of study treatment.
Groups:
- Dose Escalation: Cohort 1.6 mg/kg: Participants with HER3-positive metastatic breast cancer who received U3-1402 1.6 mg/kg administered via intravenous (IV) solution at 3-week intervals.
- Dose Escalation: Cohort 3.2 mg/kg: Participants with HER3-positive metastatic breast cancer who received U3-1402 3.2 mg/kg administered via intravenous (IV) solution at 3-week intervals.
- Dose Escalation/Dose Finding: Cohort 4.8 mg/kg: Participants with HER3-positive metastatic breast cancer who received U3-1402 4.8 mg/kg administered via intravenous (IV) solution at 3-week intervals.
- Dose Escalation/Dose Finding: Cohort 6.4 mg/kg: Participants with HER3-positive metastatic breast cancer who received U3-1402 6.4 mg/kg administered via intravenous (IV) solution at 3-week intervals.
- Dose Escalation: Cohort 8.0 mg/kg: Participants with HER3-positive metastatic breast cancer who received U3-1402 8.0 mg/kg administered via intravenous (IV) solution at 3-week intervals.
- Dose Finding: 3.2/4.8/6.4 mg/kg: Participants with HER3-positive metastatic breast cancer who received U3-1402 (Cycle 1: 3.2 mg/kg IV infusion Q3W; Cycle 2: 4.8 mg/kg IV infusion Q3W; Cycle 3 and all subsequent cycles: 6.4 mg/kg IV infusion Q3W).
- Dose Finding: 4.2/6.4 mg/kg: Participants with HER3-positive metastatic breast cancer who received U3-1402 (Cycles 1-3: 4.2 mg/kg IV infusion Q3W; Subsequent cycles: 6.4 mg/kg IV infusion Q3W).
- Dose Expansion: HER3 High 4.8 mg/kg: Participants with HER3-high, HER2-negative, HR-positive breast cancer who received 4.8 mg/kg of U3-1402 administration via intravenous (IV) solution at 3-week intervals.
- Dose Expansion: HER3-High 6.4 mg/kg: Participants with HER3-high, HER2-negative, HR-positive breast cancer who received 6.4 mg/kg of U3-1402 administration via intravenous (IV) solution at 3-week intervals.
- Dose Expansion: HER3-Low 6.4 mg/kg: Participants with HER3-low, HER2-negative, HR-positive breast cancer who received 6.4 mg/kg of U3-1402 administration via intravenous (IV) solution at 3-week intervals.
- Dose Expansion: TNBC 6.4 mg/kg: Participants with HER3-High, triple negative breast cancer who received 6.4 mg/kg of U3-1402 administration via intravenous (IV) solution at 3-week intervals.
Period: Dose Escalation
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Started | 3 | 3 | 15 | 15 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 15 | 15 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease per RECIST v1.1 | 3 | 3 | 11 | 10 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Clinical progression | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Due to side effect management of chemotherapy | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Due to investigator's decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Finding
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 12 | 12 | 0 | 0 | 0 | 0
Not completed — Progressive disease per RECIST v1.1 | 0 | 0 | 0 | 0 | 0 | 8 | 11 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Period: Dose Expansion
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 31 | 21 | 31
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 33 | 31 | 21 | 31
Not completed — Progressive disease per RECIST v1.1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 24 | 17 | 23
Not completed — Clinical progression | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3 | 1 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Not completed — Due to investigator's decision considering patient's liver condition | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Due to investigator's decision due to patient's general condition | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Due to investigator's decision because patient was a candidate for surgery | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Patient withdrew consent following 50 treatment cycles | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Groups:
- Dose Finding: 3.2/4.8/6.4 mg/kg: Participants who received U3-1402 (Cycle 1: 3.2 mg/kg IV infusion Q3W; Cycle 2: 4.8 mg/kg IV infusion Q3W; Cycle 3 and all subsequent cycles: 6.4 mg/kg IV infusion Q3W).
- Dose Finding: 4.2/6.4 mg/kg: Participants who received U3-1402 (Cycles 1-3: 4.2 mg/kg IV infusion Q3W; Subsequent cycles: 6.4 mg/kg IV infusion Q3W).
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg | Total
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6 | 12 | 12 | 33 | 31 | 21 | 31 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (10.41) | 62.3 (22.74) | 52.1 (13.38) | 58.7 (11.76) | 50.2 (8.45) | 51.8 (13.79) | 50.7 (11.92) | 56.0 (11.95) | 56.9 (11.04) | 55.4 (12.92) | 58.0 (13.73) | 55.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 15 | 15 | 6 | 12 | 12 | 33 | 31 | 21 | 31 | 182
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11 | 6 | 6 | 34
  Black of African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4
  Asian | 3 | 3 | 15 | 15 | 6 | 12 | 12 | 19 | 18 | 15 | 24 | 142
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs)
Description: AEs will be collected systematically from signing of the informed consent form (ICF) through 28 days after last dose
Time Frame: Baseline up to 28 days post last dose, up to approximately 9 months
Population: Adverse events are reported from the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6 | 12 | 12 | 33 | 31 | 21 | 31
Participants
  Any TEAE | 3 | 3 | 15 | 15 | 6 | 12 | 12 | 32 | 31 | 21 | 31
  Any TEAE Grade ≥3 | 2 | 1 | 11 | 13 | 5 | 7 | 4 | 20 | 24 | 16 | 27
  Any TEAE associated with death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 1
  Any TEAE associated with study treatment discontinuation | 0 | 0 | 1 | 2 | 2 | 3 | 0 | 4 | 2 | 1 | 3
  Any TEAE associated with dose interruption | 1 | 2 | 7 | 12 | 3 | 8 | 6 | 16 | 15 | 10 | 20
  Any TEAE associated with dose reduction | 0 | 0 | 2 | 3 | 5 | 2 | 0 | 4 | 9 | 2 | 8

2. Primary Outcome: Number of Participants With Best Overall Tumor Response Using Blinded Independent Central Review Based on Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
Description: CR was defined as a disappearance of all target and non-target lesions, PR was defined as at least a 30% decrease in the sum of diameters of target and non-target lesions, and stable disease (SD) was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD; at least a 20% increase in the sum of diameters of target and non-target lesions. Objective response rate is the number of patients with confirmed complete response and confirmed partial response.
Time Frame: From screening until disease progresses, up to approximately 9 months
Population: Best overall tumor response was assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6 | 12 | 12 | 33 | 31 | 21 | 31
Participants
  Complete response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response (PR) | 0 | 1 | 5 | 7 | 3 | 5 | 3 | 11 | 5 | 7 | 5
  Stable disease (SD)/Non-CR/Non-PD | 2 | 2 | 7 | 8 | 2 | 5 | 6 | 19 | 17 | 7 | 21
  Progressive disease (PD) | 1 | 0 | 3 | 0 | 1 | 2 | 2 | 1 | 7 | 3 | 3
  Nonevaluable (NE) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 4 | 2
  Objective response rate (ORR) | 0 | 1 | 5 | 7 | 3 | 5 | 3 | 11 | 5 | 7 | 5

3. Secondary Outcome: Dose Escalation Part: Area Under the Serum Concentration Time Curve (AUC) of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6
ng*d/mL
  AUClast, Cycle 1: number analyzed (Participants) | 3 | 3 | 12 | 11 | 6
  AUClast, Cycle 1 | 2470 (435) | 4420 (1020) | 8690 (1070) | 13000 (3310) | 16700 (4170)
  AUClast, Cycle 3: number analyzed (Participants) | 1 | 3 | 6 | 8 | 1
  AUClast, Cycle 3 | 2400 | 5920 (1070) | 13800 (3730) | 20500 (4070) | 27100
  AUCtau, Cycle 1 | 2470 (438) | 4420 (1020) | 8600 (1870) | 13600 (3020) | 16700 (4170)
  AUCtau, Cycle 3: number analyzed (Participants) | 1 | 3 | 10 | 13 | 3
  AUCtau, Cycle 3 | 2420 | 5900 (2050) | 13700 (3700) | 20300 (3200) | 21000 (5420)
  AUCinf, Cycle 1 | 2490 (440) | 4470 (1060) | 8990 (2230) | 14600 (3510) | 18300 (4920)

4. Secondary Outcome: Dose Finding Part: AUC of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 4, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg
Number analyzed (Participants) | 11 | 12
ng*d/mL
  AUClast, Cycle 1: number analyzed (Participants) | 11 | 10
  AUClast, Cycle 1 | 5540 (2020) | 7160 (1900)
  AUClast, Cycle 3: number analyzed (Participants) | 6 | 10
  AUClast, Cycle 3 | 18300 (2740) | 9360 (3670)
  AUClast, Cycle 4: number analyzed (Participants) | 0 | 8
  AUClast, Cycle 4 |  | 23100 (8130)
  AUCtau, Cycle 1 | 6160 (1160) | 7630 (1920)
  AUCtau, Cycle 3: number analyzed (Participants) | 9 | 10
  AUCtau, Cycle 3 | 16600 (3760) | 11600 (1880)
  AUCtau, Cycle 4: number analyzed (Participants) | 0 | 9
  AUCtau, Cycle 4 |  | 22300 (8010)
  AUCinf, Cycle 1 | 6220 (1200) | 7800 (1990)

5. Secondary Outcome: Dose Expansion Part: AUC of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng*d/mL
Arm/Group | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 30 | 29 | 21 | 30
ng*d/mL
  AUClast, Cycle 1: number analyzed (Participants) | 19 | 23 | 20 | 17
  AUClast, Cycle 1 | 10500 (2850) | 11500 (3930) | 11100 (4840) | 11400 (3820)
  AUClast, Cycle 3: number analyzed (Participants) | 25 | 17 | 9 | 16
  AUClast, Cycle 3 | 14200 (6540) | 20000 (14400) | 19300 (6830) | 20400 (6230)
  AUCtau, Cycle 1 | 10100 (2480) | 11900 (3400) | 11700 (4430) | 11700 (3380)
  AUCtau, Cycle 3: number analyzed (Participants) | 27 | 16 | 10 | 20
  AUCtau, Cycle 3 | 15600 (6850) | 22400 (12700) | 20300 (6830) | 19800 (5540)

6. Secondary Outcome: Dose Escalation Part: Maximum Plasma Concentration (Cmax) of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed using the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6
ng/mL
  Cmax, Cycle 1 | 1040 (217) | 1740 (421) | 2950 (661) | 3660 (1080) | 4210 (568)
  Cmax, Cycle 3: number analyzed (Participants) | 1 | 3 | 11 | 13 | 3
  Cmax, Cycle 3 | 948 | 1820 (284) | 3020 (572) | 3870 (488) | 3720 (973)

7. Secondary Outcome: Dose Finding Part: Cmax of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 4, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg
Number analyzed (Participants) | 12 | 12
ng/mL
  Cmax, Cycle 1 | 1980 (300) | 2370 (566)
  Cmax, Cycle 3: number analyzed (Participants) | 9 | 11
  Cmax, Cycle 3 | 4230 (1120) | 2830 (760)
  Cmax, Cycle 4: number analyzed (Participants) | 0 | 9
  Cmax, Cycle 4 |  | 4310 (1120)

8. Secondary Outcome: Dose Expansion Part: Cmax of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 33 | 30 | 21 | 31
ng/mL
  Cmax, Cycle 1 | 3010 (631) | 3520 (619) | 3630 (744) | 3610 (878)
  Cmax, Cycle 3: number analyzed (Participants) | 28 | 19 | 11 | 21
  Cmax, Cycle 3 | 3020 (606) | 4000 (672) | 4150 (892) | 4090 (506)

9. Secondary Outcome: Dose Escalation Part: Time to Maximum Plasma Concentration (Tmax) of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6
hours
  Tmax, Cycle 1 | 1.85 [1.80 to 1.88] | 1.68 [1.65 to 2.05] | 1.83 [1.70 to 7.13] | 2.05 [1.68 to 22.83] | 1.98 [1.77 to 6.92]
  Tmax, Cycle 3: number analyzed (Participants) | 1 | 3 | 11 | 13 | 3
  Tmax, Cycle 3 | 2.18 | 1.83 [1.83 to 2.10] | 1.88 [0.73 to 2.08] | 2.03 [0.77 to 4.13] | 4.22 [2.02 to 6.92]

10. Secondary Outcome: Dose Finding Part: Tmax of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 4, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg
Number analyzed (Participants) | 12 | 12
hours
  Tmax, Cycle 1 | 1.86 [1.60 to 4.23] | 2.01 [1.73 to 3.95]
  Tmax, Cycle 3: number analyzed (Participants) | 9 | 11
  Tmax, Cycle 3 | 2.00 [0.82 to 4.00] | 1.93 [0.60 to 3.95]
  Tmax, Cycle 4: number analyzed (Participants) | 0 | 9
  Tmax, Cycle 4 |  | 1.83 [0.73 to 6.95]

11. Secondary Outcome: Dose Expansion Part: Tmax of Anti-HER3-ac-DXd
Description: The serum concentrations for anti-HER3-ac-DXd were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 33 | 30 | 21 | 31
hours
  Tmax, Cycle 1 | 1.90 [1.72 to 7.92] | 1.97 [1.60 to 3.98] | 1.98 [1.75 to 7.50] | 1.95 [1.67 to 6.78]
  Tmax, Cycle 3: number analyzed (Participants) | 28 | 19 | 11 | 21
  Tmax, Cycle 3 | 1.78 [0.63 to 7.10] | 0.93 [0.57 to 6.80] | 2.02 [0.70 to 7.02] | 2.03 [0.77 to 6.97]

12. Secondary Outcome: Dose Escalation Part: Area Under the Concentration-Time Curve of Total Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6
ug*d/mL
  AUClast, Cycle 1: number analyzed (Participants) | 3 | 3 | 12 | 11 | 6
  AUClast, Cycle 1 | 114 (14.7) | 219 (61.0) | 416 (128) | 635 (171) | 847 (248)
  AUClast, Cycle 3: number analyzed (Participants) | 1 | 3 | 6 | 8 | 1
  AUClast, Cycle 3 | 111 | 312 (124) | 700 (234) | 1080 (280) | 1570
  AUCtau, Cycle 1 | 114 (14.5) | 219 (61.0) | 408 (115) | 671 (169) | 848 (248)
  AUCtau, Cycle 3: number analyzed (Participants) | 1 | 3 | 9 | 11 | 3
  AUCtau, Cycle 3 | 111 | 311 (122) | 682 (194) | 1050 (249) | 1200 (450)
  AUCinf, Cycle 1: number analyzed (Participants) | 3 | 3 | 15 | 13 | 4
  AUCinf, Cycle 1 | 115 (14.3) | 226 (67.3) | 447 (153) | 729 (186) | 839 (203)

13. Secondary Outcome: Dose Finding Part: Area Under the Concentration-Time Curve in Total Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 4, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg
Number analyzed (Participants) | 11 | 11
ug*d/mL
  AUClast, Cycle 1: number analyzed (Participants) | 11 | 10
  AUClast, Cycle 1 | 235 (92.7) | 302 (87.4)
  AUClast, Cycle 3: number analyzed (Participants) | 6 | 10
  AUClast, Cycle 3 | 933 (174) | 486 (199)
  AUClast, Cycle 4: number analyzed (Participants) | 0 | 8
  AUClast, Cycle 4 |  | 1110 (280)
  AUCtau, Cycle 1 | 253 (58.0) | 341 (103)
  AUCtau, Cycle 3: number analyzed (Participants) | 9 | 10
  AUCtau, Cycle 3 | 839 (220) | 616 (138)
  AUCtau, Cycle 4: number analyzed (Participants) | 0 | 9
  AUCtau, Cycle 4 |  | 1090 (276)
  AUCinf, Cycle 1: number analyzed (Participants) | 11 | 9
  AUCinf, Cycle 1 | 260 (63.4) | 335 (102)

14. Secondary Outcome: Dose Expansion Part: Area Under the Concentration-Time Curve in Total Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug*d/mL
Arm/Group | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 31 | 26 | 20 | 30
ug*d/mL
  AUClast, Cycle 1: number analyzed (Participants) | 19 | 24 | 20 | 17
  AUClast, Cycle 1 | 525 (174) | 570 (248) | 543 (225) | 528 (166)
  AUClast, Cycle 3: number analyzed (Participants) | 25 | 17 | 9 | 16
  AUClast, Cycle 3 | 831 (391) | 1070 (656) | 1070 (381) | 1000 (266)
  AUCtau, Cycle 1 | 483 (140) | 564 (178) | 580 (200) | 542 (158)
  AUCtau, Cycle 3: number analyzed (Participants) | 25 | 16 | 10 | 19
  AUCtau, Cycle 3 | 874 (365) | 1200 (536) | 1030 (366) | 940 (243)

15. Secondary Outcome: Dose Escalation Part: Cmax of Total Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were assessed in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6
ug/mL
  Cmax, Cycle 1 | 39.8 (9.55) | 61.6 (8.41) | 95.8 (13.5) | 136 (26.8) | 149 (35.3)
  Cmax, Cycle 3: number analyzed (Participants) | 1 | 3 | 11 | 13 | 3
  Cmax, Cycle 3 | 37.6 | 66.8 (11.2) | 112 (14.1) | 149 (24.7) | 165 (25.4)

16. Secondary Outcome: Dose Finding Part: Cmax of Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 4, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg
Number analyzed (Participants) | 12 | 12
ug/mL
  Cmax, Cycle 1 | 67.9 (11.3) | 87.2 (33.2)
  Cmax, Cycle 3: number analyzed (Participants) | 9 | 11
  Cmax, Cycle 3 | 139 (25.0) | 94.9 (10.6)
  Cmax, Cycle 4: number analyzed (Participants) | 0 | 9
  Cmax, Cycle 4 |  | 145 (16.6)

17. Secondary Outcome: Dose Expansion Part: Cmax in Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 33 | 30 | 21 | 31
ug/mL
  Cmax, Cycle 1 | 107 (20.3) | 129 (21.2) | 126 (28.4) | 127 (24.4)
  Cmax, Cycle 3: number analyzed (Participants) | 28 | 19 | 11 | 21
  Cmax, Cycle 3 | 121 (27.7) | 152 (25.8) | 140 (29.7) | 146 (21.7)

18. Secondary Outcome: Dose Escalation Part: Tmax of Total Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were assessed in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg
Number analyzed (Participants) | 3 | 3 | 15 | 15 | 6
hours
  Tmax, Cycle 1 | 1.85 [1.80 to 2.17] | 1.68 [1.65 to 1.70] | 1.95 [1.70 to 6.87] | 2.00 [1.82 to 7.00] | 2.14 [1.77 to 6.92]
  Tmax, Cycle 3: number analyzed (Participants) | 1 | 3 | 11 | 13 | 3
  Tmax, Cycle 3 | 2.18 | 1.83 [1.83 to 2.10] | 1.88 [0.67 to 6.88] | 2.02 [0.75 to 96.42] | 2.07 [2.02 to 2.13]

19. Secondary Outcome: Dose Finding Part: Tmax of Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 4, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were analyzed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg
Number analyzed (Participants) | 12 | 12
hours
  Tmax, Cycle 1 | 1.85 [1.60 to 4.07] | 1.80 [1.73 to 6.83]
  Tmax, Cycle 3: number analyzed (Participants) | 9 | 11
  Tmax, Cycle 3 | 3.80 [0.75 to 6.97] | 1.93 [0.65 to 4.07]
  Tmax, Cycle 4: number analyzed (Participants) | 0 | 9
  Tmax, Cycle 4 |  | 3.80 [0.67 to 4.10]

20. Secondary Outcome: Dose Expansion Part: Tmax in Anti-HER3 Antibody
Description: The serum concentrations for total anti-HER3 antibody LC/MS were quantified using the IC-LC/MS assay.
Time Frame: Cycle 1, Day 1 to Cycle 3, Day 21 (each cycle is 21 days)
Population: Pharmacokinetic data were assessed in participants with available data in the Pharmacokinetic Analysis Set.
Measure: Median (Full Range); unit: hours
Arm/Group | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
Number analyzed (Participants) | 33 | 30 | 21 | 31
hours
  Tmax, Cycle 1 | 1.92 [1.75 to 6.80] | 2.00 [1.60 to 4.13] | 1.87 [1.75 to 6.80] | 1.93 [1.67 to 22.02]
  Tmax, Cycle 3: number analyzed (Participants) | 28 | 19 | 11 | 21
  Tmax, Cycle 3 | 1.95 [0.68 to 6.97] | 2.10 [0.73 to 7.17] | 1.98 [0.73 to 6.98] | 2.00 [0.65 to 6.90]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline up to 28 days post last dose, up to 9 months.
Arm/Group | Dose Escalation: Cohort 1.6 mg/kg | Dose Escalation: Cohort 3.2 mg/kg | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg | Dose Escalation: Cohort 8.0 mg/kg | Dose Finding: 3.2/4.8/6.4 mg/kg | Dose Finding: 4.2/6.4 mg/kg | Dose Expansion: HER3 High 4.8 mg/kg | Dose Expansion: HER3-High 6.4 mg/kg | Dose Expansion: HER3-Low 6.4 mg/kg | Dose Expansion: TNBC 6.4 mg/kg
All-Cause Mortality (participants affected / at risk) | 2/3 | 2/3 | 13/15 | 11/15 | 2/6 | 10/12 | 10/12 | 22/33 | 24/31 | 18/21 | 16/31
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 3/15 | 9/15 | 2/6 | 4/12 | 3/12 | 10/33 | 12/31 | 7/21 | 8/31
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 15/15 | 15/15 | 6/6 | 12/12 | 12/12 | 32/33 | 31/31 | 21/21 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Cohort 1.6 mg/kg (N=3) | Dose Escalation: Cohort 3.2 mg/kg (N=3) | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg (N=15) | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg (N=15) | Dose Escalation: Cohort 8.0 mg/kg (N=6) | Dose Finding: 3.2/4.8/6.4 mg/kg (N=12) | Dose Finding: 4.2/6.4 mg/kg (N=12) | Dose Expansion: HER3 High 4.8 mg/kg (N=33) | Dose Expansion: HER3-High 6.4 mg/kg (N=31) | Dose Expansion: HER3-Low 6.4 mg/kg (N=21) | Dose Expansion: TNBC 6.4 mg/kg (N=31)
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 3 | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Delirum (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: Cohort 1.6 mg/kg (N=3) | Dose Escalation: Cohort 3.2 mg/kg (N=3) | Dose Escalation/Dose Finding: Cohort 4.8 mg/kg (N=15) | Dose Escalation/Dose Finding: Cohort 6.4 mg/kg (N=15) | Dose Escalation: Cohort 8.0 mg/kg (N=6) | Dose Finding: 3.2/4.8/6.4 mg/kg (N=12) | Dose Finding: 4.2/6.4 mg/kg (N=12) | Dose Expansion: HER3 High 4.8 mg/kg (N=33) | Dose Expansion: HER3-High 6.4 mg/kg (N=31) | Dose Expansion: HER3-Low 6.4 mg/kg (N=21) | Dose Expansion: TNBC 6.4 mg/kg (N=31)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 6 | 4 | 0 | 3 | 3 | 5 | 3 | 5 | 3
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 3 | 1 | 1 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 3 | 2
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 8 | 8 | 3 | 4 | 1 | 13 | 19 | 5 | 10
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 4 | 8 | 4 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 4 | 8 | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Iodine allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergy to arthropod sting (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 9 | 11 | 4 | 5 | 4 | 18 | 15 | 8 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 2 | 1 | 4 | 0 | 8 | 3 | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 3 | 0 | 0 | 1 | 6 | 5 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 5 | 2 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 4 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 4 | 1 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 3 | 2 | 0 | 4 | 1 | 6 | 3 | 1 | 4
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 5 | 0 | 2 | 2 | 2 | 1 | 1 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 4 | 3 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 2 | 0 | 1 | 1 | 2 | 1 | 2 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 3 | 4 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Punctate keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival deposit (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 6 | 1 | 0 | 2 | 4 | 5 | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 1 | 1 | 2 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 11 | 14 | 6 | 12 | 10 | 22 | 25 | 15 | 25
Vomiting (Gastrointestinal disorders) | 2 | 2 | 8 | 9 | 4 | 4 | 3 | 15 | 13 | 7 | 17
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 5 | 8 | 1 | 5 | 6 | 15 | 14 | 7 | 14
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 6 | 7 | 2 | 2 | 2 | 6 | 5 | 10 | 12
Constipation (Gastrointestinal disorders) | 1 | 0 | 3 | 5 | 3 | 4 | 1 | 8 | 11 | 6 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 2 | 2 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 2 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Angular cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 5 | 4 | 1 | 0 | 7 | 9 | 6 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 5 | 0 | 1 | 1 | 4 | 1 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 2 | 3 | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 1 | 1 | 1 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin sensitisation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 4 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5 | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Pubic pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 5 | 5 | 2 | 5 | 2 | 10 | 10 | 8 | 10
Malaise (General disorders) | 0 | 0 | 2 | 8 | 2 | 2 | 3 | 9 | 5 | 3 | 10
Pyrexia (General disorders) | 1 | 0 | 2 | 3 | 1 | 1 | 2 | 5 | 6 | 4 | 4
Oedema peripheral (General disorders) | 0 | 0 | 1 | 5 | 0 | 0 | 0 | 3 | 2 | 1 | 1
Pain (General disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 10 | 13 | 3 | 4 | 4 | 15 | 13 | 11 | 17
Neutrophil count decreased (Investigations) | 0 | 0 | 10 | 13 | 2 | 8 | 3 | 15 | 10 | 8 | 15
White blood cell count decreased (Investigations) | 0 | 0 | 9 | 14 | 2 | 6 | 2 | 12 | 10 | 7 | 10
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 10 | 7 | 3 | 3 | 1 | 11 | 11 | 6 | 10
Alanine aminotransferase increased (Investigations) | 1 | 0 | 9 | 4 | 3 | 2 | 1 | 11 | 10 | 7 | 10
Weight decreased (Investigations) | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 8 | 7 | 1 | 3
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3 | 3 | 1 | 2 | 0 | 1 | 5 | 2 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 4 | 1 | 2 | 0 | 6 | 3 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 2 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 3 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intraocular pressure increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood electrolytes decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body in eye (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation fibrosis - lung (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 2 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Corneal disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Peripheral sweling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT02980341/Prot_SAP_000.pdf